CLINICAL TRIAL: NCT00915980
Title: Meal Stimulating After Roux-en Y Gastric Bypass
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Collaborators: University of Copenhagen (Other); Novo Nordisk A/S (Industry)
Responsible Party: Siv Hesse Jacobsen, MD, Hvidovre University Hospital
Other Study IDs: H-C-2007-0108
Record Dates: First submitted 2009-06-05; First posted 2009-06-08 (Estimated); Last update posted 2011-07-08 (Estimated); Status verified 2011-07

CONDITIONS: Gastric Bypass; Obesity
Keywords: Meal-test; reduced OGTT; gastric bypass surgery and glucose metabolism; Glucose metabolism before and after gastric bypass; Different OGTT; New meal- test
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma and serum sampels for analysis of primarily intestinal hormones
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients without diabetes undergoing gastric bypass
  Interventions: Procedure: gastric bypass surgery and testing

INTERVENTIONS:
Procedure: gastric bypass surgery and testing — The patients will be tested with OGTT and meal testing before and after undergoing gastric bypass surgery.

SUMMARY:
In many studies, gastric bypass surgery led to total remission of type 2 diabetes (T2DM) as early as 1 - 2 days after surgery before any real weight loss has occurred. This suggests that the remission of the T2DM is due to the direct effect of the operation, more than the secondary effect of the weight loss. The reasons for the major effect on the glucose metabolism after gastric bypass surgery are still unaccounted for.

The aim of this project will be to unveil some of the mechanisms that explain the effect of gastric bypass surgery on the glucose metabolism. Further more to find a better way of testing patients that have just undergone gastric bypass surgery. It is not possible to test patients who have just undergone gastric bypass surgery with normal oral glucose tolerance test (OGTT) and a normal meal, because patients can only take in fluid and a normal OGTT will often lead to dumping. Instead we will try to modify these tests - OGTT with lower glucose level and meal-testing with a protein drink.

The hypothesis of the study is that the investigators can see changes in different hormones and adipokines before and after surgery, even with modified OGTT and meal testing. The project will consist of clinical trials on patients without T2DM that will undergo gastric bypass surgery. The studies will take place before and within the first week after surgery. The investigators will measure different hormones and adipokines after OGTT and a meal with a protein drink. The investigators expect to see significant changes in some of the analyses after the operation in patients undergoing gastric bypass.

ELIGIBILITY:
Inclusion Criteria:

* Obese with BMI> 40 undergoing gastric bypass surgery OR
* Obese with BMI > 35 with complications of their obesity in form of high blood pressure or other related complications undergoing gastric bypass surgery
* Age between 20-60 years

Exclusion Criteria:

* Age > 60
* Diabetes
* Psychiatric illness
* Mentally challenged
* Addiction
* Serious cardiac or lung diseases
* Diseases in the abdomen
* Other serious illness

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Obese with BMI > 40 undergoing gastric bypass surgery or obese with BMI > 35 with complications of their obesity in form of high blood pressure or other related complications undergoing gastric bypass surgery.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2008-01; Primary Completion 2009-05 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre hospital, Hvidovre, Denmark